CLINICAL TRIAL: NCT04461457
Title: Targeted Radiation Therapy for Ovarian Cancer: Intraperitoneal Treatment With 211-astatine-MX35 F(ab')2
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Swedish Cancer Society (Other); The Swedish Research Council (Other Government); Sahlgrenska University Hospital (Other)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 001-211Astatine; 151:2004/26262 (Other: Swedish Medical Products Agency (MPA)); S571-03 (Other: Ethics committee, Sahlgrenska Academy, Göteborg University)
Record Dates: First submitted 2020-06-29; First posted 2020-07-08 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Intervention Model Description: To investigate the pharmacokinetics of the conjugate 211At-MX35 F(ab') 2.
  Groups of 3 patients will be treated at increasing activity concentrations starting at 50 MBq/L
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intraperitoneal Radioimmunotherapy boost (Experimental): Four groups of 3 patients with recurring ovarian cancer treated by salvage chemo-therapy and being in complete or good partial remission will receive one IP dose of 211astatine-MX35 F(ab'2). Starting at 50 MBq/L. Dose escalation 100 Mbq/L, 200 MBq/L and finally 300 MBq/L.
  Interventions: Combination Product: 211-astatine MX35 F(ab')2

INTERVENTIONS:
Combination Product: 211-astatine MX35 F(ab')2 — Alpha emitting radionuclide 211At conjugated to monoclonal antibody MX35 F(ab')2. Targeting the sodium phosphate transporter (NaPi2b).

SUMMARY:
In this alpha-radioimmunotherapy study groups of 3 patients with recurring epithelial ovarian cancer treated by salvage chemo-therapy and being in complete or good partial remission will receive one intra peritoneal infusion of 211 astatine (211At)-MX35 F(ab')2 . Patients will receive a single dose of MX35 F(ab')2 radiolabeled with increasing activity concentration of 211At in 1.0 - 2 L Extraneal® solution starting at an activity concentration of 50 megabecquerel per litre (MBq/L).

DETAILED DESCRIPTION:
* Five days prior to therapy the patient is provided with a central intra venous line and an abdominal catheter will be introduced during laparoscopy. To investigate the access to the whole abdominal cavity and possible catheter leakage, a 99mTc-colloid, will be infused intra peritoneally (IP) within 1.0 L of a gluco-polymer (Extraneal®).
* At the day of treatment vital signs will be measured prior to and after the 30 min infusion and at least every second hour during the first 6 hours after infusion, daily for the remainder of the in-hospital stay and at a minimum at 2, 3, 4 and 8 weeks after the IP infusion. Blood samples will be obtained for pharmacokinetic analyses every hour after completion of the IP infusion for 8 hours, then every 6 hours, together with sampling from the i.p. catheter.
* SPECT imaging of the whole abdominal cavity and thorax including the thyroid may be performed following completion of the IP infusion and at approx 8 or 20hrs post infusion.
* Physical examination and electrocardiogram will be done prior to and 4 weeks after the IP infusion. Clinical biochemical and hematological parameters will be monitored weekly after treatment. Blood samples to evaluate immunogenicity as well as cancer antigen-125 (CA-125) will also be taken at 2 and 8 weeks after treatment.
* The first patient will be observed for at least 4 weeks with any observed toxicity is Grade 2 or less, before the additional patient is accrued at the dose level.
* Dosimetry safety criteria: Based upon published data on maximal tolerated absorbed dose (Gy) recalculated to equivalent dose (Sv) with the assumption that the relative biological effectiveness (RBE) = 5, a limit for organ doses is defined. If any organ would reach the defined limit the study will be stopped.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically confirmed ovarian or tubal or primary peritoneal adenocarcinoma.
2. Patients must have a recurrent intraperitoneal cancer and treated by a salvage chemotherapy to complete or good partial remission
3. The following laboratory and clinical results within 2 weeks prior to first study day:

   Absolute neutrophil count (ANC) > 1.5 x 109/L Platelet count > 100 x 109/L Serum bilirubin < upper limit of normal(ULN) Aspartate aminotransaminase (ASAT) < 1.5 x ULN Serum aminotransferase (ALAT) < 1.5 x ULN Serum creatinine < 1.5 x upper limit of normal Thyreoglobulin baseline information Thyroid-stimulating hormone (TSH) baseline information T4 baseline information
4. Karnofsky performance status > 70.
5. Must understand written and spoken Swedish
6. Before any trial-specific procedures or treatment can be performed, the patient must give written informed consent for participation in the trial.

Exclusion Criteria:

1. Active parenchymal disease (distant metastasis) (i.e. stage IV International Federation of Gynecology and Obstetrics (FIGO) classification.
2. Presence of diagnosed extra abdominal metastasis
3. Clinically significant heart disease.
4. Electrocardiographic demonstrating clinically significant arrhythmias.
5. Other serious illnesses, e.g. serious infections requiring antibiotics, coagulation disorders.
6. Chronic inflammatory bowel disease.
7. Chemotherapy, biologic therapy, or immunotherapy within 4 weeks prior
8. Advanced abdominal adherences.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2005-02-05 (Actual); Primary Completion 2011-03-19 (Actual); Study Completion 2012-01-19 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration (Cmax) of Astatine 211 | Sampled from +1 hour to +48 hrs post infusion.
  Decay corrected activity concentration in serum, intraperitoneal fluid and urine.
Area under the curve (AUC) of astatine 211 from time of dosing to 48 hrs after dosing | Sampled from +1 hour to +48 hrs post infusion.
  Decay corrected activity concentration in serum, intraperitoneal fluid and urine, including actual imaging quantification on gamma-Camera scintigraphy.
Toxicity: hematology, liver, kidney, thyroid function | From procedure start (implantation of catheter) to 8 weeks after infusion
  As defined by NCI Common Toxicity Criteria v2.0

CONTACTS AND LOCATIONS:
Locations (1):
- Sahlgrenska University Hospital, Dept of Oncology, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No
Upun specific request, data could be considered to be shared.

REFERENCES:
- [Result] Andersson H, Cederkrantz E, Back T, Divgi C, Elgqvist J, Himmelman J, Horvath G, Jacobsson L, Jensen H, Lindegren S, Palm S, Hultborn R. Intraperitoneal alpha-particle radioimmunotherapy of ovarian cancer patients: pharmacokinetics and dosimetry of (211)At-MX35 F(ab')2--a phase I study. J Nucl Med. 2009 Jul;50(7):1153-60. doi: 10.2967/jnumed.109.062604. Epub 2009 Jun 12. PMID 19525452
- [Result] Cederkrantz E, Andersson H, Bernhardt P, Back T, Hultborn R, Jacobsson L, Jensen H, Lindegren S, Ljungberg M, Magnander T, Palm S, Albertsson P. Absorbed Doses and Risk Estimates of (211)At-MX35 F(ab')2 in Intraperitoneal Therapy of Ovarian Cancer Patients. Int J Radiat Oncol Biol Phys. 2015 Nov 1;93(3):569-76. doi: 10.1016/j.ijrobp.2015.07.005. Epub 2015 Jul 11. PMID 26460999
- [Result] Hallqvist A, Bergmark K, Back T, Andersson H, Dahm-Kahler P, Johansson M, Lindegren S, Jensen H, Jacobsson L, Hultborn R, Palm S, Albertsson P. Intraperitoneal alpha-Emitting Radioimmunotherapy with 211At in Relapsed Ovarian Cancer: Long-Term Follow-up with Individual Absorbed Dose Estimations. J Nucl Med. 2019 Aug;60(8):1073-1079. doi: 10.2967/jnumed.118.220384. Epub 2019 Jan 25. PMID 30683761